CLINICAL TRIAL: NCT06444646
Title: The Adipose Tissue and Sex-specific Role of Adipose-derived Extracellular Vesicles in Obesity-related Skeletal Muscle Insulin Resistance.
Brief Title: Differences in Extracellular Vesicles From Adipose Tissue of Individuals With Obesity.
Acronym: EVO
Status: Recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Research Foundation Flanders (Other); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, prof. dr. Kenneth Verboven, Prof. dr., Hasselt University
Other Study IDs: CTU Z-2022041
Record Dates: First submitted 2023-02-27; First posted 2024-06-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood + subcutaneous/visceral adipose tissue biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EVO participants with obesity: From each patient, two adipose tissue biopsies will be taken during bariatric surgery; one from the subcutaneous and one from the visceral adipose tissue.
  Interventions: Other: Adipose tissue biopsy; Other: Blood sampling; Other: Questionnaire; Other: Patient phenotyping
- EVO participants without obesity: From each lean patient, two adipose tissue biopsies will be taken during abdominal surgery; one from the subcutaneous and one from the visceral adipose tissue.
  Interventions: Other: Adipose tissue biopsy; Other: Blood sampling; Other: Questionnaire; Other: Patient phenotyping

INTERVENTIONS:
Other: Adipose tissue biopsy — From each patient, two biopsies will be taken during surgery; one from the subcutaneous and one from the visceral adipose tissue.
Other: Blood sampling — From each patient, two venous blood samples (citrate, LiHe and EDTA plasma) will be taken before surgery.
Other: Questionnaire — Before bariatric surgery, every patient will fill out questions about general health (physical activity, sedentary behavior, sleeping pattern, ...), physical condition before surgery (nausea, food intake, ...), etc.
Other: Patient phenotyping — Length and weight will be measured to calculate body mass index (BMI). Waist and hip circumference will be assessed, as well as blood pressure (both systolic and diastolic) and heart rate at rest. Body composition will be determined using a bioelectrical impedance analysis (BIA) in the hospital. Medication use and comorbidities (that are allowed within the in-/exclusion criteria) will also be derived from the patient's medical files with patient's permission.

SUMMARY:
Our society is characterized by a strong increase in the prevalence of obesity, which often causes the development of cardiovascular and metabolic diseases such as type 2 diabetes. The way(s) obesity is responsible for these diseases, is still insufficiently understood. This study therefore examines the content of human fat tissue storage location- and cell type-specific extracellular vesicles (EVs) in lean and obese individuals, and the possible connection with sex, insulin sensitivity, and the blood-brain barrier.

DETAILED DESCRIPTION:
This study focuses on unraveling the fundamental differences in communication via extracellular vesicles (EVs) derived from fat cells and immune cells in terms of fat tissue storage location and sex among individuals with and without obesity. The study hypothesizes that the differences in EV profiles, originating from corresponding in vitro differentiated hMADS and ex vivo isolated adult fat cells and immune cells, among individuals with and without obesity can be related to sex and/or fat tissue storage location. Additionally, the effect of the isolated EVs on the blood-brain barrier function is also investigated.

ELIGIBILITY:
Individuals with obesity - Inclusion Criteria:

* Caucasian adults with obesity that have a body mass index (BMI) of at least 35 kg/m^2 and are scheduled for their first bariatric surgery.
* Final male/female ratio of this study is 1:1
* Minimal knowledge of Dutch to read and understand the informed consent.

Individuals with obesity - Exclusion Criteria:

* Smoking and/or drug abuse
* Cardiovascular diseases (including but not limited to implanted aids like a pacemaker or defibrillator)
* Lung and/or kidney diseases
* Brain and/or nerve diseases
* Malignant diseases (e.g. cancer)

Individuals without obesity (lean) - inclusion criteria

* Caucasian adults with obesity that have a body mass index (BMI) of between 18 and 24.9 kg/m^2 and are scheduled for abdominal surgery
* Female only
* Minimal knowledge of Dutch to read and understand the informed consent.

Individuals without obesity (lean) - exclusion criteria

* Smoking and/or drug abuse
* Cardiovascular diseases (including but not limited to implanted aids like a pacemaker or defibrillator)
* Lung and/or kidney diseases
* Brain and/or nerve diseases
* Endocrine diseases like type 2 diabetes
* Malignant diseases (e.g. cancer)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with or without obesity presenting at the bariatric surgery or abdominal surgery department, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
General characterization of adipocyte- or adipose tissue-derived extracellular vesicles | Baseline
  Concentration, size, surface markers, content and morphology of extracellular vesicles derived from isolated mature adipocytes, isolated adipose tissue stem cells or isolated from complete adipose tissue explants derived from both the subcutaneous as the visceral adipose tissue biopsies will be investigated.
General characterization of adipose tissue- and blood immune cells | Baseline
  Immune cells isolated from adipose tissue and blood will be characterized by flow cytometry.

OTHER OUTCOMES:
Correlations between possible influencing patient factors (derived by a questionnaire) and extracellular vesicle characteristics | Baseline
  Questions about general health (physical activity, sedentary behavior, sleeping pattern, ...), physical condition before surgery (nausea, food intake, ...), etc. This information will be used to make correlations with extracellular vesicles characteristics.
Correlations between possible influencing patient factors (derived by patient phenotyping) and extracellular vesicle characteristics | Baseline
  Length and weight will be measured to calculate body mass index (BMI). Waist and hip circumference will be assessed, as well as blood pressure (both systolic and diastolic) and heart rate at rest. Body composition will be determined using a bioelectrical impedance analysis (BIA). Medicine use and comorbidities (that are allowed within the in-/exclusion criteria) will also be derived from the patient's medical files with patient's permission. This information will be used to make correlations with extracellular vesicles characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No
Patient information will be coded based on unique identifiers. This file will only be available for the principle investigator and will be stored safely on the secured Google Enterprise drive of UHasselt. Biological samples will be processed and coded by UHasselt, after registration in the biobank of Limburg (UBILIM). Only researchers of the EVO study will have access to any of the files, patient information or biological samples.